CLINICAL TRIAL: NCT06608407
Title: The Effect of Platelet Rich Plasma in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Brief Title: Platelet Rich Plasma in the Prevention of Adhesion Reformation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Yang Ling Ling, Dr, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024FXHEC-KSP020
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-09

CONDITIONS: Intrauterine Adhesion; Asherman Syndrome
Keywords: intrauterine adhesion; platelet rich plasma; hysteroscopic adhesiolysis; Fertility outcome
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP Group (Experimental): After the completion of hysteroscopic adhesiolysis, recruited participants will be randomized to one of the two treatment groups by computer-generated numbers: Immediately administer uterine perfusion with PRP after surgery, and administered PRP perfusion during hysteroscopy at 4 and 8 weeks after hysteroscopic adhesiolysis, A second-look hysteroscopy and ultrasound assessment of the endometrium will be carried out 4 weeks after the surgery, and again at 8 weeks after the surgery.
  Interventions: Biological: PRP group
- Control group (No Intervention): Control group without PRP treatment.

INTERVENTIONS:
Biological: PRP group — After the completion of hysteroscopic adhesiolysis, recruited participants will be randomized to one of the two treatment groups by computer-generated numbers: Immediately administer uterine perfusion with PRP after surgery, and administered PRP perfusion during hysteroscopy at 4 and 8 weeks after hysteroscopic adhesiolysis, A second-look hysteroscopy and ultrasound assessment of the endometrium will be carried out 4 weeks after the surgery, and again at 8 weeks after the surgery. Control group without PRP treatment.
  Arms: PRP Group

SUMMARY:
Asherman syndrome, which occurs after trauma to the basalis layer of the endometrium. It seems that the role of postoperative platelet rich plasma（PRP）therapy in the prevention of recurrence of IUA is still controversial. To investigate if PRP therapy can prevent adhesion reformation after adhesiolysis.

After the completion of hysteroscopic adhesiolysis, recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: having PRP after hysteroscopic adhesiolysis; and the control group without PRP treatment. A second-look hysteroscopy and ultrasound assessment of the endometrium will be carried out 4 weeks after the surgery, and again at 8 weeks after the surgery.

DETAILED DESCRIPTION:
Asherman syndrome, which occurs after trauma to the basalis layer of the endometrium. It seems that the role of postoperative platelet rich plasma（PRP）therapy in the prevention of recurrence of IUA is still controversial. To investigate if PRP therapy can prevent adhesion reformation after adhesiolysis.

After the completion of hysteroscopic adhesiolysis, recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: having PRP after hysteroscopic adhesiolysis; and the control group without PRP treatment. A second-look hysteroscopy and ultrasound assessment of the endometrium will be carried out 4 weeks after the surgery, and again at 8 weeks after the surgery.

Background information Asherman syndrome, which occurs after trauma to the basalis layer of the endometrium generally after endometrial curettage, may manifest as hypomenorrhea, amenorrhea, dysmenorrhea, infertility or recurrent miscarriage.

At present, hysteroscopic adhesiolysis is the recommended standard diagnostic method and treatment for IUA. Recurrence of uterine cavity adhesion post-operatively is frequently reported, especially in severe IUA patients. A number of strategies have been proposed to prevent recurrence of adhesion reformation, including the use of post-operative PRP. However, it is still not known if PRP therapy is indeed necessary or effective. In a prospective randomized study which evaluated the efficacy of PRP in preventing IUA following hysteroscopic adhesiolysis , it was found that PRP did not have any benefit in reducing adhesion formation. In another RCT study on women with Asherman syndrome, there did not appear to be any difference in the recurrence of IUA and pregnancy rate between those who did or did not receive PRP medication. It seems that the role of postoperative PRP therapy in the prevention of recurrence of IUA is still controversial. In this prospective, randomized, controlled study, the investigators wish to determine if PRP therapy is of benefit in preventing adhesion reformation after IUA for Asherman syndrome. As the effect may be different for subjects with different degrees of IUA, the investigators propose to stratify the subjects into those with mild and severe IUAs.

Objectives To investigate if PRP therapy can prevent adhesion reformation after adhesiolysis.

Participants The participants will be recruited from the hysteroscopy Center of the Fuxing Hospital, Beijing, China. Before the surgery all patients with suspected Asherman syndrome will undergo preoperative evaluations, including a detailed history of the menstrual pattern, any previous intrauterine surgery, reproductive history, as well as trans-vaginal ultrasonography. The severity and extent of intrauterine adhesions will be scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version). The inclusion criteria include women aged 18-40 years; written consent obtained; and agreement to have second-look hysteroscopy. The exclusion criteria included:1. has received estrogen therapy within 3 month of enrolment. 2. suffers from leiomyoma, endometrial polyps, cancer, or polycystic ovarian syndrome (PCOS). 3.History of genital tuberculosis.

Study Design After the completion of hysteroscopic adhesiolysis, recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: Immediately administer uterine perfusion with PRP after surgery, and administered PRP perfusion during hysteroscopy at 4 and 8 weeks after hysteroscopic adhesiolysis, A second-look hysteroscopy and ultrasound assessment of the endometrium will be carried out 4 weeks after the surgery, and again at 8 weeks after the surgery. Power Calculation On the basis of the results of the comparing previous research on using PRP to prevent IUA recurrence, the estimated IUA recurrence rates in subjects with moderate to severe IUA (AFS score 7-12) are 25% in the PRP group and 54% in the control group. Accepting a type 1 error (a) of 0.05, and a type 2 error (b) of 0.10, the number of subjects in each arm of the randomized, controlled trial would be 41. Assuming that the dropout rate is 10%, the total number of subject to be recruited would be 46 in each arm. the total number of subject to be recruited would be 46 in each arm. Procedure Surgical procedure The surgery will be carried out by one of three experienced hysteroscopic surgeons with the use of a 4.5-mm rigid hysteroscope (Olympus) with 5% saline perfusion under 100 mm Hg pressure. The primary procedure will be performed under general anesthesia in a day surgery unit. Ultrasonographic guidance will be routinely used. Once the extent and severity of uterine adhesion has been assessed, the adhesions will be divided with the use of mono-polar instrument until normal uterine anatomy is achieved.

Postoperative treatments All subjects will be treated with oral antibiotic for 5 days. Second-look hysteroscopy will be carried out in the early proliferative phase, 4 weeks after the initial operation; a third-look hysteroscopy will be carried out 8 weeks after the initial operation. After assessment of the extent and severity of any reformed adhesion, hysteroscopic adhesiolysis will be carried out at the time of the second-look or third-look procedure, if adhesion had recurred. The surgeon who later performs the second-look and third-look hysteroscopy will be blinded to the randomization.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Asherman's syndrome. AFS score >7.

Exclusion Criteria:

1. Leiomyoma;
2. Endometrial polyps;
3. Ppolycystic ovarian syndrome (PCOS).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
AFS Score at Third-look Hysteroscopy | 8 weeks after operation
  The investigators measured the AFS score between the PRP group and Control group through hysteroscopy 8 weeks after operation. American Fertility Society [(AFS) score in intrauterine adhesion who underwent hysteroscopic adhesiolysis.The higher the score, the heavier the degree of adhesion.
  The AFS (American Fertility Society) scoring system for endometrial assessment is as follows:
  Extent of involvement: 1 point(<1/3 of the uterine cavity); 2 points(1/3 to 2/3 of the uterine cavity); 4 points(2/3 of the uterine cavity).
  Type of adhesion:1 point(Filmy); 2 points(Filmy and dense); 4 points(Dense) . Menstrual pattern:1 point(Normal menses); 2 points(Menstrual reduction); 4 points(Amenorrhea) .
  Points are summed to give a total score ranging from 1 to 12, which is used to classify the degree of endometrial injury or disease:Mild (Grade I): 1 to 4 points;Moderate (Grade II): 5 to 8 points;Severe (Grade III): 9 to 12 points.
Endometrial thickness under ovulation ultrasound | 3 months
  Ultrasound measurement of endometrial thickness during ovulation period three months after adhesion release surgery

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fu Xing Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fuxing hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No